CLINICAL TRIAL: NCT03407157
Title: Oral Probiotic Supplementation in Pregnancy to Reduce Group B Streptococcus Colonization
Acronym: OPSiP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Dublin City University (Other)
Responsible Party: Principal Investigator, Michelle Butler, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H17-02189
Record Dates: First submitted 2017-12-07; First posted 2018-01-23 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Group B Streptococcus Carrier in Childbirth
Keywords: Probiotics; Pregnancy; GBS; Group B Streptococcus

STUDY DESIGN:
Intervention Model Description: Randomisation will be centrally controlled using iSTAR, a web-based computerised randomisation platform at the BC Children's Hospital Research Institute, run by the PRE-EMPT (Pre-eclampsia Eclampsia Monitoring Prevention and Treatment) research group, UBC. PRE-EMPT will provide the randomisation platform, and web-linked drug supply management system. Randomisation will occur in random blocks of 2 and 4. Women will be randomised on a 1:1 ratio to probiotic:placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomisation process will assign each participant with a unique study ID number. This study ID number will be required when allocating study drug bottles and lozenge packages and for recording data on the case report form (CRF). The drug bottle number and lozenge packs will be dispensed by a study team member directly to the participant. Probiotics and placebos will look and taste identical and drug bottles and lozenge packs and labels will look identical.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Probiotic supplementation
  Interventions: Dietary Supplement: Probiotic supplementation
- Control (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic supplementation — Participants will take two capsules daily of Urex Plus VCap-5 (each containing 2.5 billion CFUs of L. rhamnosus and L. reuteri) and one lozenge of Blis K12 (1 billion CFUs of streptococcus Salivarius)
  Arms: Intervention
Other: Placebo — Participants will be asked to take 2 placebo capsules and 1 placebo lozenge daily from 25 weeks pregnancy
  Arms: Control

SUMMARY:
This is a double-blind randomized placebo controlled trial that will investigate whether the use of three specific species of probiotics taken orally in pregnancy from 25 weeks gestation will reduce the incidence of Group B Streptococcus (GBS) colonization. Participants will take 2 capsules and 1 lozenge per day of either probiotic or placebo from 25 weeks gestation. The primary outcome will be the study-specific vaginal/rectal swab collected after 35 weeks gestation and before delivery. A reduction in women testing positive for GBS would lead to a decrease risk to infants of GBS infection and a reduction in the use of antibiotics leading to less maternal and neonatal antibiotic exposure.

DETAILED DESCRIPTION:
Background:

Group B streptococcus (GBS) infection of the newborn is a leading cause of neonatal morbidity and mortality in North America. Up to 30% of pregnant women are colonized with GBS. Half of the babies born to colonized mothers will become colonized themselves, and of those, about 1-2% may develop early onset GBS infection (EOGBS), which is associated with significant mortality (between 5% and 20%) and morbidity (71% bacteremia, 11% meningitis, 19% pneumonia). The current recommendation is for routine administration of IPA to women who test positive for GBS at term. Although IPA therapy may reduce the incidence of neonatal GBS infection, it can increase the risk of other infections such as E. Coli, neonatal thrush, and ampicillin resistant Enterobacteriaceae.

There is also accumulating evidence linking antibiotics in pregnancy with childhood asthma, childhood obesity, and obesity in later life. IPA is also associated with antibiotic resistance, diarrhoea (including Clostridium difficile), and fungal infections. There is a growing worldwide interest in utilizing probiotics to enhance and manipulate the human microbiome in order to reduce a wide range of communicable and non-communicable diseases. Probiotics have been studied extensively in pregnant women and are considered safe and well tolerated when ingested or used vaginally.

Probiotics in pregnancy may reduce GBS colonization and the need for intrapartum antibiotic prophylaxis through a number of mechanisms. Some probiotics produce antibacterial substances and film-like barriers to pathogens. By adhering to vaginal epithelial cells, probiotics also displace pathogens such as GBS. S. salivarius K12 has been shown to inhibit several GBS strains, including disease-implicated isolates from newborns and colonizing isolates from the vaginal tract of pregnant women. In vivo and in vitro studies demonstrate its ability to adhere to the vaginal epithelium and directly impair the growth and adherence of GBS.

Several pilot randomized trials of L. reuteri and L. rhamnosus show promise in their their ability to reduce GBS colonization and have been shown to be safe. In vivo and in vitro studies of various lactobacillus strains, including rhamnosus and reuteri, have demonstrated an inhibitory effect on GBS.

Preliminary research to date suggests the administration of probiotic supplements to women in pregnancy may reduce the incidence of GBS colonization, thus reducing the need to administer intravenous prophylactic antibiotics (IPA) to women during labour. The specific species of probiotics chosen for this trial create a combination of inhibitory and antibacterial effects that may result in a greater reduction of GBS colonization than shown in previous trials.

The study:

The OPSiP study is a three-year, two-centre, double blind randomized placebo controlled trial. The aim of this study is to assess if a combined daily oral supplementation of Lactobacillus rhamnosus, Lactobacillus reuteri and Streptococcus salivarius beginning from 25 weeks gestation and continued until delivery will reduce vaginal/rectal group B streptococcus (GBS) colonization rates. Secondary aims include reduction of maternal and neonatal antibiotic exposure, and maternal vaginal and urinary tract infections.

450 healthy pregnant women receiving care from a regulated maternity care professional and registered at either St. Paul's or BC Women's Hospitals in Vancouver, British Columbia will be recruited. Women will be introduced to the study through posters and flyers and information from their maternity care provider. Women will be provided with verbal and written information on the study and provide written consent to participate before being entered into the study. Women will be entered into the study following initial screening to confirm their eligibility to participate in the study and then randomized to the intervention or control group.

Women randomized to the intervention group will receive a daily combination of one lozenge and two capsules of oral probiotic supplements comprised of three probiotic species; Lactobacillus rhamnosus and Lactobacillus reuteri (Urex Plus VCap-5) and Streptococcus salivarius K12 (Blis K12). The control arm will receive identical placebos administered using the same route and regimen as the active probiotic. Both groups will begin taking their daily study lozenges and capsules at 25 weeks gestation until delivery.

Five study-specific swabs will be collected, three vaginal/rectal and two oral swabs. The first vaginal/rectal swab and the first oral swab will be obtained at intake, after randomization and prior to the start of the intervention. The second vaginal/rectal swab will be obtained at mid-point, between 29-33 weeks gestational age. The third vaginal/rectal swab and second oral swab will be collected between 35 weeks and delivery.

The primary outcome will be vaginal/rectal GBS status, ascertained from the last study-specific vaginal/rectal swab. Statistical analysis will be on the basis of intention to treat. Treatment effect will be estimated using logistic regression. A two-tailed p-value <0.05 will be considered significant.

Secondary analysis will be performed on last observation moving forward, protocol-compliant groups and with adjustment for care-provider type and use of other dietary probiotic sources.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with a singleton
* Gestational age between 23 and 25+0 weeks
* Over the age of 18
* Registered for delivery, at one of the participating centres
* Under the care of a regulated maternity care provider (midwife, obstetrician (OB), or family physician).

Exclusion Criteria:

* Unable to provide consent
* Fetus has known major anomalies
* Significant immunosuppression
* Type I or Type II diabetes (non-gestational)
* Previous infant with GBS (these women will automatically be advised to be treated with IV antibiotic therapy)
* GBS bacteriuria diagnosed in present pregnancy (reasoning as per above)
* Plans to use oral or vaginal probiotic supplementation/therapy (capsules/tablets/lozenges/drinks) during their pregnancy (outside of natural food sources; yogurt, kimchi, kombucha etc)
* Enrolled in another study that involves the administration of a drug/product

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 168 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be vaginal/rectal GBS colonization status at delivery | Last vaginal/rectal swab taken after 35 weeks gestation and prior to delivery
  Measured using the study-specific rectal/vaginal swab

SECONDARY OUTCOMES:
Maternal antibiotic exposure | Questionnaires administered at intake (22-25 weeks), mid-term (29-33 weeks), term (35-37 weeks) and chart review (6 weeks post-birth)
  Women will be asked in each questionnaire if they have had any antibiotics prescribed and if so for the name of the antibiotic. Information will also be collected on antibiotics prescribed from medical records
Maternal urinary tract infections | Questionnaires administered at intake (22-25 weeks), mid-term (29-33 weeks), term (35-37 weeks) and chart review (6 weeks post-birth)
  Women will be asked in each questionnaire if they have been diagnosed with a urinary tract infection and if so, if antibiotics were prescribed. Information will also be collected from medical records
Maternal bacterial vaginosis infections | Questionnaires administered at intake (22-25 weeks), mid-term (29-33 weeks), term (35-37 weeks) and chart review (6 weeks post-birth)
  Women will be asked in each questionnaire if they have been diagnosed with bacterial vaginosis and if so, if treatment was prescribed. Information will also be collected from medical records
Maternal vaginal candida infections | Questionnaires administered at intake (22-25 weeks), mid-term (29-33 weeks), term (35-37 weeks) and chart review (4-6 weeks postpartum)
  Women will be asked in each questionnaire if they have been diagnosed with vaginal candida (yeast) infection and if so, if treatment was prescribed. Information will also be collected from medical records

OTHER OUTCOMES:
Passage of probiotic strains to gastrointestinal tract and vaginal epithelium and adherence | Oral and vaginal/rectal swabs taken at 23-25 weeks, 29-33 weeks, and 35 weeks
  Presence of three probiotic strains (L. rhamnosus GR-1, L. reuteri RC-14, and S. salivarius K12) in swabs taken over the course of the study
Adverse events | From the time of randomisation to 28 days of discontinuing the study supplements
  From health care provider notification, participant notification, semi-weekly chart audits, participant questionnaires
Gestational diabetes | Number of Participants with gestational diabetes recorded in chart review at 4-6 weeks postpartum
  Recorded in medical records
Pre-term labour | Number of Participants with pre-term labour, recorded in chart review at 4-6 weeks postpartum
  Recorded in medical records
Pre-term and pre-labour rupture of membranes | Number of Participants with pre-term and pre-labour rupture of membranes, recorded in chart review at 4-6 weeks postpartum
  Recorded in medical records
Chorio-amnionitis | Number of Participants with chorio-amnionities, recorded in chart review at 4-6 weeks postpartum
  Recorded in medical records
Maternal BMI | Chart review at 4-6 weeks postpartum
  Recorded in medical records
Pre- and/or post-partum depression | Number of Participants with pre- and/or post-partum depression, recorded in chart review at 4-6 weeks postpartum
  Any diagnosis of pre- and/or post-partum depression, date of onset, duration and treatment prescribed recorded in medical records.
Infant birth weight | Chart review at 4-6 weeks postpartum
  Recorded in medical records
Infant APGAR scores at 1, 5 and 10 minutes after birth | Chart review at 4-6 weeks postpartum
  As recorded in medical records
(Direct) infant exposure to antibiotics | Chart review at 4-6 weeks postpartum
  Recorded in medical records
Admission of infant to Neonatal Intensive Care Unit (NICU) | Chart review at 4-6 weeks postpartum
  Recorded in medical records
Early onset neonatal infections, including GBS | Chart review at 4-6 weeks postpartum
  Recorded in medical records

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Butler, PhD, RM, Principal Investigator — Dublin City University; Patricia Janssen, PhD, Principal Investigator — UBC School of Population and Public Health
Locations (2):
- Canada (2):
  - BC Women's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
Pending approval from the REC and once all final results have been published, de-identified data will be made available upon request for secondary use of data. Any proposed projects for secondary use must be approved by the study working group and the local REB.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After primary trial results have been accepted for publication
Access Criteria: Access criteria are de-identified data only and requires approval as stated above from the trial working group and local REB

REFERENCES:
- [Background] Bizzarro MJ, Dembry LM, Baltimore RS, Gallagher PG. Changing patterns in neonatal Escherichia coli sepsis and ampicillin resistance in the era of intrapartum antibiotic prophylaxis. Pediatrics. 2008 Apr;121(4):689-96. doi: 10.1542/peds.2007-2171. PMID 18381532
- [Background] Cox LM, Blaser MJ. Antibiotics in early life and obesity. Nat Rev Endocrinol. 2015 Mar;11(3):182-90. doi: 10.1038/nrendo.2014.210. Epub 2014 Dec 9. PMID 25488483
- [Background] de Vrese M. Health benefits of probiotics and prebiotics in women. Menopause Int. 2009 Mar;15(1):35-40. doi: 10.1258/mi.2009.009008. PMID 19237621
- [Background] Glasgow TS, Young PC, Wallin J, Kwok C, Stoddard G, Firth S, Samore M, Byington CL. Association of intrapartum antibiotic exposure and late-onset serious bacterial infections in infants. Pediatrics. 2005 Sep;116(3):696-702. doi: 10.1542/peds.2004-2421. PMID 16140710
- [Background] Hanson L, Vandevusse L, Duster M, Warrack S, Safdar N. Feasibility of oral prenatal probiotics against maternal group B Streptococcus vaginal and rectal colonization. J Obstet Gynecol Neonatal Nurs. 2014 May-Jun;43(3):294-304. doi: 10.1111/1552-6909.12308. Epub 2014 Apr 22. PMID 24754328
- [Background] Elias J, Bozzo P, Einarson A. Are probiotics safe for use during pregnancy and lactation? Can Fam Physician. 2011 Mar;57(3):299-301. PMID 21402964
- [Background] Money D, Allen VM; INFECTIOUS DISEASES COMMITTEE. The prevention of early-onset neonatal group B streptococcal disease. J Obstet Gynaecol Can. 2013 Oct;35(10):939-948. doi: 10.1016/S1701-2163(15)30818-5. PMID 24165063
- [Background] Mueller NT, Whyatt R, Hoepner L, Oberfield S, Dominguez-Bello MG, Widen EM, Hassoun A, Perera F, Rundle A. Prenatal exposure to antibiotics, cesarean section and risk of childhood obesity. Int J Obes (Lond). 2015 Apr;39(4):665-70. doi: 10.1038/ijo.2014.180. Epub 2014 Oct 9. PMID 25298276
- [Background] Ohlsson A, Shah VS. Intrapartum antibiotics for known maternal Group B streptococcal colonization. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD007467. doi: 10.1002/14651858.CD007467.pub3. PMID 23440815
- [Background] PHAC (2011) Steptococcus Agalactiae, Pathogen Safety Data Sheet. Public Health Agency of Canada. Available at: http://www.phac-aspc.gc.ca/lab-bio/res/psds-ftss/streptococcus-agalactiae-eng.php
- [Background] Stensballe LG, Simonsen J, Jensen SM, Bonnelykke K, Bisgaard H. Use of antibiotics during pregnancy increases the risk of asthma in early childhood. J Pediatr. 2013 Apr;162(4):832-838.e3. doi: 10.1016/j.jpeds.2012.09.049. Epub 2012 Nov 6. PMID 23140881
- [Background] Juarez Tomas MS, Ocana VS, Nader-Macias ME. Viability of vaginal probiotic lactobacilli during refrigerated and frozen storage. Anaerobe. 2004 Feb;10(1):1-5. doi: 10.1016/j.anaerobe.2004.01.002. PMID 16701493
- [Background] Reid G. Probiotic and prebiotic applications for vaginal health. J AOAC Int. 2012 Jan-Feb;95(1):31-4. doi: 10.5740/jaoacint.sge_reid. PMID 22468339
- [Background] Kaewsrichan J, Peeyananjarassri K, Kongprasertkit J. Selection and identification of anaerobic lactobacilli producing inhibitory compounds against vaginal pathogens. FEMS Immunol Med Microbiol. 2006 Oct;48(1):75-83. doi: 10.1111/j.1574-695X.2006.00124.x. PMID 16965354
- [Background] Ortiz L, Ruiz F, Pascual L, Barberis L. Effect of two probiotic strains of Lactobacillus on in vitro adherence of Listeria monocytogenes, Streptococcus agalactiae, and Staphylococcus aureus to vaginal epithelial cells. Curr Microbiol. 2014 Jun;68(6):679-84. doi: 10.1007/s00284-014-0524-9. Epub 2014 Jan 28. PMID 24469557
- [Background] Pascual LM, Daniele MB, Ruiz F, Giordano W, Pajaro C, Barberis L. Lactobacillus rhamnosus L60, a potential probiotic isolated from the human vagina. J Gen Appl Microbiol. 2008 Jun;54(3):141-8. doi: 10.2323/jgam.54.141. PMID 18654035
- [Background] Patras KA, Wescombe PA, Rosler B, Hale JD, Tagg JR, Doran KS. Streptococcus salivarius K12 Limits Group B Streptococcus Vaginal Colonization. Infect Immun. 2015 Sep;83(9):3438-44. doi: 10.1128/IAI.00409-15. Epub 2015 Jun 15. PMID 26077762
- [Background] Ho M, Chang YY, Chang WC, Lin HC, Wang MH, Lin WC, Chiu TH. Oral Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 to reduce Group B Streptococcus colonization in pregnant women: A randomized controlled trial. Taiwan J Obstet Gynecol. 2016 Aug;55(4):515-8. doi: 10.1016/j.tjog.2016.06.003. PMID 27590374
- [Background] Wickens KL, Barthow CA, Murphy R, Abels PR, Maude RM, Stone PR, Mitchell EA, Stanley TV, Purdie GL, Kang JM, Hood FE, Rowden JL, Barnes PK, Fitzharris PF, Crane J. Early pregnancy probiotic supplementation with Lactobacillus rhamnosus HN001 may reduce the prevalence of gestational diabetes mellitus: a randomised controlled trial. Br J Nutr. 2017 Mar;117(6):804-813. doi: 10.1017/S0007114517000289. Epub 2017 Apr 3. PMID 28367765
- [Background] Di Pierro F, Colombo M, Zanvit A, Risso P, Rottoli AS. Use of Streptococcus salivarius K12 in the prevention of streptococcal and viral pharyngotonsillitis in children. Drug Healthc Patient Saf. 2014 Feb 13;6:15-20. doi: 10.2147/DHPS.S59665. eCollection 2014. PMID 24600248
- [Background] Acikgoz ZC, Gamberzade S, Gocer S, Ceylan P. [Inhibitor effect of vaginal lactobacilli on group B streptococci]. Mikrobiyol Bul. 2005 Jan;39(1):17-23. Turkish. PMID 15900833
- [Derived] Hayes K, Janssen P, Payne BA, Jevitt C, Johnston W, Johnson P, Butler M. Oral Probiotic Supplementation in Pregnancy to Reduce Group B Streptococcus Colonisation (OPSiP trial): study protocol for a double-blind parallel group randomised placebo trial. BMJ Open. 2024 Feb 5;14(2):e076455. doi: 10.1136/bmjopen-2023-076455. PMID 38316588